CLINICAL TRIAL: NCT00348452
Title: Double-blind, Randomized, Dose-ranging, Parallel-group Comparison of the Efficacy and Safety of Extended Release Tramadol Hydrochloride (Tramadol HCl ER) 100 mg, 200 mg, 300 mg, Celecoxib 200 mg and Placebo in the Treatment of Osteoarthritis of the Knee and/or Hip.
Brief Title: A Study Comparing the Effectiveness and Safety of Extended Release Tramadol HCl at 100 mg, 200 mg and 300 mg Doses to Placebo for the Treatment of Moderate to Severe Pain Due to Osteoarthritis (OA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B02.CT3.021.TRA P03
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Pain
Keywords: osteoarthritis pain; knee; hip; extended release analgesia; opioid
MeSH Terms: conditions — Chronic Pain | interventions — Celecoxib

INTERVENTIONS:
Drug: tramadol HCl ER; celecoxib

SUMMARY:
The purpose of this study is to compare the analgesic efficacy and safety of tramadol HCl ER 100 mg, 200 mg and 300 mg once a day (QD), with placebo in patients with moderate to severe pain due to OA. For the purposes of this study, celecoxib will serve as a positive control to validate the sensitivity of the model. The study hypothesis is that tramadol HCl ER is safe and effective in the treatment of moderate to severe pain due to OA.

DETAILED DESCRIPTION:
Immediate release (IR) tramadol has demonstrated efficacy in several pain conditions including, obstetrical, gynecological, orthopedic, abdominal, and oral surgery. The short elimination half-life of IR tramadol necessitates every 4-6 hour dosing to maintain optimum levels of analgesia in chronic pain. The study medication in this study is a once-daily, extended release (ER) tramadol formulation. This is a 12-week multicenter, double-blind, randomized, dose-ranging, placebo and positive-controlled, parallel-group study. For the purpose of this study, celecoxib serves as a positive control to validate the sensitivity of the model. Patients with OA functional Class I-III of the knee or hip, with moderate to severe pain are eligible for participation, if appropriate criteria are met. During a 2-7 day washout period, the use of all analgesic medications will be discontinued. Eligible patients experiencing moderate to severe pain (>= 40 mm on a 100 mm visual analog scale) in the index joint to be evaluated and who meet all other study criteria will enter the double-blind titration period. During this period, patients will be randomly assigned to receive treatment with tramadol HCl ER 100 mg, 200 mg, 300 mg, celecoxib 200 mg or placebo, once daily. During the titration period (Days 1-9) all patients will be contacted by phone every few days to ensure they do not experience unmanageable pain or unacceptable side effects. Efficacy and safety evaluations will be collected at study visits occurring at Weeks 1, 2, 3, 6, 9 and 12 or at the time of early termination. Study medication will be discontinued at Week 12 and patients will return after 1 week for a post-treatment visit (Week 13).

ELIGIBILITY:
Inclusion Criteria:

* Patients with American College of Rheumatology (ACR) Functional Class I-III OA of the knee or hip;
* Patients with involvement of knee or hip joint that warrants treatment with COX-2 selective inhibitors, NSAIDs, acetaminophen, or opioid analgesics for at least 75 of the 90 days preceding the screening visit;
* Patients with a pain intensity score in index joint >= 40 mm on the visual analog scale(VAS) at the baseline visit;
* Patients who are able to discontinue acetaminophen, NSAIDS, COX-2 selective inhibitors and other analgesics during the washout period and all analgesics other than the study medication throughout the study;
* Patients who are able to understand the study procedures and complete the pain scales.

Exclusion Criteria:

* Patients with a medical condition, other than OA, uncontrolled with treatment or any clinically significant condition that, in the investigator's opinion, precludes study participation or interferes with the assessment of chronic pain and other OA symptoms;
* Patients with a diagnoses of inflammatory arthritis, gout, pseudo-gout or Paget's disease, that, in the investigator's opinion, interferes with the assessment of pain and other symptoms of OA;
* Patients with a diagnosis of chronic pain syndrome;
* Patients with an ACR or a clinical diagnosis of fibromyalgia;
* Patients with any other clinically significant form of joint disease or prior joint replacement surgery at the index joint;
* Patients with an anticipated need for surgery or other invasive procedure in the index joint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-09; Study Completion 2003-08

PRIMARY OUTCOMES:
The primary outcome is the change from baseline to week 12 in the WOMAC OA Index pain and physical function subscale scores and the patient global assessment of disease activity.

SECONDARY OUTCOMES:
The secondary outcomes include: change from baseline in the daily arthritis pain intensity scores from patient diaries, WOMAC OA stiffness subscale scores, OA pain intensity VAS for index and non-index joints, and Chronic Pain Sleep Inventory scale